CLINICAL TRIAL: NCT03005470
Title: Technology for Innovative Monitoring of Cardiovascular Prevention: A Precision Randomized Controlled Trial
Brief Title: Technology for Innovative Monitoring of Cardiovascular Prevention: a RCT
Acronym: TIM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Sandra Costa Fuchs, Professor Sandra C. Fuchs, MD, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 31423214.0.0000.5327
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Blood Pressure, High; Prehypertension
Keywords: Prehypertension; Hypertension; Blood pressure; Intervention; Lifestyle; Blood pressure monitoring; Ambulatory Blood Pressure Monitoring; Text Messages; High blood pressure
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Intervention Model Description: This is a factorial randomized controlled trial (Figure 1) of effectiveness of the use of technologies - smartphones and blood pressure monitoring - to reduce systolic blood pressure and change lifestyle.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants have uncontrolled hypertension under on pharmacological treatment. They will be requested not to change drugs and medicine doses during the trial.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TELEM group (Experimental): Participants in the telemonitoring home blood pressure group will receive an oscillometric monitor to measure blood pressure at home for six months. Measurements will be made for at least five days a week (including one day during the weekend). Each blood pressure measure will be sent to the center of the study coordination center through software downloaded on the participant's smartphone.
  Interventions: Device: TELEM
- TELEMEV group (Experimental): In the telemonitoring of lifestyle group, participants will receive customized standardized text messages to stimulate lifestyle changes and adherence to blood pressure lowering medication. The messages will be focused on the adoption of DASH diet, sodium restriction, increase of physical activity, weight control and adherence to drug treatment. They will be sent to the smarphones on four of the five days of the week at random times using a software developed for this study.
  Interventions: Device: TELEMEV
- TELEM-TELEMEV group (Experimental): Participants in the telemonitoring home blood pressure plus telemonitoring of lifestyle group (TELEM-TELEMEV) will receive both interventions as previously described.
  Interventions: Device: TELEM-TELEMEV
- Usual clinical treatment (UCT) (Active Comparator): Participants in the control group will be under antihypertensive treatment, chosen at the discretion of the assistant physician. Participants will not receive any technological tool to stimulate blood pressure control or lifestyle modification.
  Interventions: Other: UCT

INTERVENTIONS:
Device: TELEM — Participants in the telemonitoring home blood pressure (TELEM) group will receive an oscillometric monitor to measure blood pressure at home for six months. Measurements will be made early in the morning (5:00 to 10:00) and in the evening (18:00 to 21:00) for at least five days a week (including one day during the weekend). Each blood pressure measure will be sent to the center of the study coordination center through software downloaded on the participant's smartphone.
  Arms: TELEM group
Device: TELEMEV — In the lifestyle telemonitoring group (TELEMEV), participants will receive customized standardized text messages to stimulate lifestyle changes and adherence to blood pressure lowering medication. The messages will be focused on the adoption of DASH diet, sodium restriction, increase of physical activity, weight control and adherence to drug treatment. They will be sent out on four of the five days of the week at random times. The messages will be sent to the smarphones through a software developed for this study.
  Arms: TELEMEV group
Device: TELEM-TELEMEV — Participants in the TELEM plus TELEMEV (TELEM-TELEMEV) will receive both interventions as previously described.
  Arms: TELEM-TELEMEV group
Other: UCT — Participants in the control group will receive usual clinical treatment (UCT) on pre-scheduled visits, but will not receive any technological tool to stimulate blood pressure control or lifestyle modification.
  Arms: Usual clinical treatment (UCT)

SUMMARY:
National and international guidelines that guide evidence-based clinical practice advocate an effort to improve blood pressure control based on changing lifestyle and use of blood pressure lowering medication. However, the effectiveness of the approach usually depends on patient adherence to both types of interventions - pharmacological and behavioral. Lack of success on blood pressure control has increased the scope of interventions to improve adherence and to reduce cardiovascular risk factors without overburdening the public health system. The use of technologies - mobile or smart phones, games, blogs, internet and video conferencing - to implement interventions can reduce costs and increase coverage.

Interactive interventions have been associated with a reduction in systolic blood pressure of 3-8 mmHg in patients with hypertension. These interventions were individually tailored to patient specificities and involved self-monitoring of blood pressure and lifestyle changes, including regular physical activity, DASH diet, restriction of dietary salt intake, and weight control. However, the effectiviness of these interventions may have short half-lives without periodic reinforcement, either to adhere to pharmacological treatment or behavioral changes. Innovative technologies can be used to achieve lasting effect and even greater blood pressure reduction.

Therefore, the purpose of this study is to compare effectiveness of four strategies to reduce blood pressure and improve lifestyle.

DETAILED DESCRIPTION:
This is a factorial randomized controlled trial of comparative effectiveness and precision medicine. Participants will be randomly assigned in a ratio of 1:1:2:1 to one of four arms: telemonitoring of blood pressure by smart phone, text message for lifestyle changes, both interventions (telemonitoring and messages) or usual clinical care. At randomization, all participants will receive a printed booklet with lifestyle modification guidelines. The standardized recommendation to adhere to the pharmacological treatment prescribed by the attending physician will also be implemented. These types of interventions do not allow the research assistant responsible for monitoring to be blinded, but the researcher resposible for the assessment of the outcome will be blinded to the allocated arm and the results will be evaluated through objective measurements.

ELIGIBILITY:
Inclusion Criteria:

* Office blood pressure: systolic blood pressure greater or equal to 135 mmHg and below 180 mmHg or diastolic blood pressure greater or equal to 85 mmhg and below 110 mmhg
* Ambulatory Blood Pressure Monitoring (ABPM): 24h-SBP ≥130 mmHg or 24h-DBP ≥80 mmHg
* Use of one or two blood pressure lowering drugs
* Have a smartphone

Exclusion Criteria:

* Cardiovascular event in the last 6 months (eg myocardial infarction, stroke, pacemaker or other use)
* Life threatening conditions, low life expectancy
* Inability to measure blood pressure;
* Previous diagnosis of secondary hypertension;
* IF WOMAN: lactating, pregnancy or who intend to become pregnant within the next 6 months.
* Unable to understand the interventions

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2017-01; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring (ABPM) | Change at six months (end of the trial)
  Reduction in 24h-systolic blood pressure

SECONDARY OUTCOMES:
ABPM | Change at six months (end of the trial)
  Reduction in 24h-diastolic blood pressure
Other ABPM measurements | Change from baseline to end of the trial
  Reduction in daytime and nighttime systolic blood pressure
Office blood pressure | At six months (end of the trial)
  Office blood pressure control rate: <130/80 mmHg
Reduction in sodium urinary excretion | Change at six months (end of the trial)
  Reduction in sodium urinary excretion in a urinary spot
Improvement of lifestyle: increase of regular physical activity, intake of DASH-type diet, or weight reduction | Change at six months (end of the trial)
  Increase in average steps taken during 7 days, using pedometer; reported dietary intake using 24h recall of food groups; reduction of reported intake, using a quantitative questionnaire; or reduction of at least 3 kg or the average reduction

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Fuchs, Principal Investigator — HCPA, UFRGS
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] David CN, Iochpe C, Harzheim E, Sesin GP, Goncalves MR, Moreira LB, Fuchs FD, Fuchs SC. Effect of Mobile Health Interventions on Lifestyle and Anthropometric Characteristics of Uncontrolled Hypertensive Participants: Secondary Analyses of a Randomized Controlled Trial. Healthcare (Basel). 2023 Apr 8;11(8):1069. doi: 10.3390/healthcare11081069. PMID 37107903
- [Derived] Fuchs SC, Harzheim E, Iochpe C, David CN, Goncalves MR, Sesin GP, Costa CM, Moreira LB, Fuchs FD. Technologies for Innovative Monitoring to Reduce Blood Pressure and Change Lifestyle Using Mobile Phones in Adult and Elderly Populations (TIM Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Aug 7;7(8):e169. doi: 10.2196/resprot.9619. PMID 30087093